CLINICAL TRIAL: NCT06698224
Title: Paired Spinal Cord and Peripheral Nerve Stimulation for Hand Function Recovery in Humans Post Cervical SCI
Brief Title: Paired Spinal Cord and Peripheral Nerve Stimulation to Recover Hand Function in SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Pawan Sharma, PT. Ph.D., Postdoctoral Fellow, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1176828
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury; Spinal Cord Disease; Spinal Cord Injuries (SCI)
Keywords: Spinal cord injury; Hand function; Spinal cord stimulation; Paired stimulation; Physical therapy
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- scTS (Active Comparator): This arm will receive 20 sessions of spinal cord transcutaneous stimulation (scTS) combined with physical therapy.
  Interventions: Device: Spinal cord transcutaneous stimulation
- scTS+PNS (Experimental): This arm will receive 20 sessions of paired application of spinal cord transcutaneous stimulation (scTS) and peripheral nerve stimulation (PNS) followed by scTS combined with physical therapy.
  Interventions: Device: Paired spinal cord and peripheral nerve stimulation

INTERVENTIONS:
Device: Spinal cord transcutaneous stimulation — Physical therapy combined with spinal cord transcutaneous stimulation will increase activity in the paralyzed or weak arm and hand muscles in individuals with spinal cord injury. Transcutaneous spinal cord stimulation is a non-invasive stimulation strategy and are known to facilitate recovery of lost function post spinal cord injury.
  Arms: scTS
Device: Paired spinal cord and peripheral nerve stimulation — Physical therapy combined with paired spinal cord-peripheral nerve stimulation will increase activity in the paralyzed or weak arm and hand muscles in individuals with spinal cord injury. Transcutaneous spinal cord and peripheral nerve stimulation are both non-invasive stimulation strategy and are known to facilitate recovery of lost function post spinal cord injury.
  Other Names: Spinal cord transcutaneous stimulation; Peripheral nerve stimulation
  Arms: scTS+PNS

SUMMARY:
Individuals who suffer a spinal cord injury in the neck region have difficulty using their hands due to paralysis and/or weakness of their arms and hand muscles. This project aims to test the effects of pairing spinal cord and nerve stimulation combined with physical therapy training in recovering arms and hand function. The long-term goal is to provide better therapies that will improve the ability of individuals with spinal cord injuries to use their arms and hands to perform everyday tasks, similar to injury before.

DETAILED DESCRIPTION:
Cervical spinal cord injury (SCI) results in paralysis and/or weakness of arms and hands that severely affects the independence and quality of life post-injury. Therefore, regaining arm and hand function remains the top priority of this population. Considering that SCI is mostly incomplete in nature, recent evidence suggests that physical or occupational therapy training combined with spinal cord transcutaneous stimulation (scTS) is effective in restoring arm and hand function post-cervical SCI. scTS is a non-invasive painless technique that augments the intrinsic capacity of the spinal cord to facilitate motor function post-SCI. The beneficial effects of scTS can be further improved by coupling it with peripheral nerve stimulation (PNS), which supplies the arm and hand muscles.

This study aims to investigate how precisely timed paired application of spinal cord transcutaneous stimulation (scTS) and peripheral nerve stimulation (PNS) combined with physical therapy can improve the use of arms and hands in those with a SCI. Spinal cord transcutaneous stimulation (scTS) is a non-invasive electrical stimulation provided on top of the skin over specific areas of the spinal cord to excite the nervous system for the activity being trained and promote connections between the brain and spinal cord. Peripheral nerve stimulation (PNS) is a non-invasive electrical stimulation provided on top of the skin over specific areas of the arm, forearm, and hand to excite the peripheral nerves and promote connections between the spinal cord and the muscles involved in the activity-based recovery training. We hypothesize that precisely timed application of scTS and PNS will increase spinal cord excitability. Increased spinal cord excitability coupled with physical therapy will facilitate hand function recovery post-SCI.

Study aims:

1. To establish optimal time sequencing for the paired scTS and PNS delivery resulting in the spinal cord motor neuron excitability in non-injured (NI) and SCI participants.
2. To investigate the acute effects of paired scTS and PNS delivery on spinal cord motor neuron and corticospinal excitability.
3. To investigate the effectiveness of paired scTS and PNS along with scTS combined with AB-UET in recovering hand function post cervical SCI.
4. To identify the potential mechanisms of action underlying the observed changes in the hand function following training with paired scTS and PNS along with scTS combined with AB-UET.

This is a pretest-posttest experimental design. SCI participants will be enrolled for Aims 1, 2, 3 and 4. For SCI participants, On site medical evaluation, ASIA Impairment Scale (ISNCSCI-AIS), MVC grip strength and nerve intactness study will be collected or performed during the screening process. If the individual is potentially eligible for the study, as determined by the study physician and investigators, they will undergo pre-training assessments, 20 training sessions, and post-training assessments. Non-Injured (NI) participants will be enrolled for Aims 1 and 2.

ELIGIBILITY:
For SCI participants:

Inclusion Criteria:

* At least 18 years of age
* Non-progressive cervical SCI
* Greater than or equal to 6-months post spinal cord injury
* Stable medical condition
* Viable median and ulnar nerve as evident from MMR and M-Wave recordings
* Wrist extensor and finger flexors score between 1-3 for both upper extremity for ISNCSCI motor assessment.

Exclusion Criteria:

* Ventilator Dependent
* Untreated fracture or pressure ulcer
* Untreated psychiatric disorder or ongoing drug abuse
* Cardiac, respiratory, bladder, renal, or other untreated medical disorder unrelated to SCI
* Skeletal muscle Botox injections less than 6 months prior
* Previous tendon transfer of the arm or arms
* Any implanted pump (i.e., baclofen pump, pain pump, etc.) prior to randomization
* Pregnant at the time of enrollment or planning to become pregnant during the course of the study
* Unable or unwilling to wean from anti-spasticity medications
* History of seizure or epilepsy
* Metal in Head
* Cochlear implant
* Implanted brain stimulators
* Aneurysm clips
* Increased intracranial pressure (which lowers seizure threshold)
* Cardiac pacemaker
* Personal or family history of epilepsy
* Tricyclic antidepressants or neuroleptics (which lower seizure threshold)

For healthy volunteer/participants:

Inclusion Criteria:

* At least 18 years of age

Exclusion Criteria:

* Neurological injury or disease
* Pregnant at the time of enrollment or planning to become pregnant during the course of the study
* Personal or family history of seizure or epilepsy
* Tricyclic antidepressants or neuroleptics (which lower seizure threshold)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
GRASSP | From enrollment to the end of treatment at 4 weeks
  Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) is a 3-part assessment designed to measure participant's hand and arm function. The test specifically measures strength, sensation, and prehension. During strength testing, selected upper extremity muscles are assessed for the grade of muscle contraction or power of the muscle. During sensation testing, specific zones on the palmar and dorsal aspects of the hand are tested with Semmes Weinstein Monofilaments (SWM) with varying weights. Prehension is assessed both qualitatively and quantitatively. During the qualitative section, no specific position is required, except that the hand should be positioned appropriately for movement with assistance from the examiner, if necessary. During quantitative section, participant is asked to perform six tasks and performance is graded.
NRS | From enrollment to the end of treatment at 4 weeks
  Neuromuscular Recovery Scale Assessment (NRS) assesses the level of muscle activation and amount of external assistance required to perform motor tasks involving hand, arm, and trunk. The research participant will be asked to perform motor tasks as independently as possible. Research staff will score each of these tasks based on the algorithm. NRS consists of six sub-items focusing on UE function, including overhead press, shoulder flexion, grasp, door pull, open with key, and can open and manipulation. Items are scored from phase 1 to phase 4, the higher the phase, the better is the functional performance
Voluntary hand opening and closing kinematics | From enrollment to the end of treatment at 4 weeks
  Three-dimensional kinematic data will be collected using a motion capture system. Reflective markers will be placed on the participant's forearm, hand, and fingers to track wrist and finger movements during a maximum hand opening and closing task. Surface electrodes will be applied on the participant's skin to acquire EMG data.
Maximal voluntary grip strength | From enrollment to the end of treatment at 4 weeks
  For maximal voluntary grip strength, participants will be instructed to apply as much force as possible while trying to grasp or making a fist around the grip handle during a 3 second audio cue. Each MVC attempt will be followed by a rest period of 20 seconds of no activity. A total of 5 grip strength attempts will be collected.
Transcranial magnetic stimulation motor evoked potential (MEP) | From enrollment to the end of treatment at 4 weeks
  To obtain MEP, transcortical magnetic stimulation (TMS) will be delivered through a figure-of-eight coil using a monophasic current waveform to the optimal scalp position along the arm and hand representation of the primary motor cortex eliciting largest MEP (MEPmax) from targeted arm and hand muscles. Electromyographic (EMG) sensors will be applied on the participant's skin to acquire muscle data.
F-wave | From enrollment to the end of treatment at 4 weeks
  120% of the maximum stimulation intensity causing plateauing of the M-wave will be used to elicit F-wave. Evoked responses will be recorded using low-noise, pre-amplified surface EMG electrodes placed on the arm and hand muscles to record signals.

SECONDARY OUTCOMES:
Functional Neurophysiological assessment (FNPA) | From enrollment to the end of treatment at 4 weeks
  The assessment will be performed with the participant in lying position. The participants will be asked to relax for a minimum of 5 minutes at the beginning of the assessment to acquire a baseline of the electrical noise in his/her muscles and in the room. Corresponding volitional motor tasks will then be performed to match the muscles being recorded at that time (elbow flexion to record from biceps brachii). Reflexive testing, including deep tendon reflexes, clonus, Babinski, and reaction to vibration may be performed after volitional testing.
Multisegmental Motor Response (MMR) | From enrollment to the end of treatment at 4 weeks
  MMR will be evoked transcutaneously by using a constant current stimulator between the C2 spinous processes and the coccyx. The cathode(s) (pre-gelled, soft surface electrodes) will be placed over the skin between C2 spinous processes and the coccyx, while large anode(s) will be placed over the clavicle, abdomen, iliac bone or at different levels or at segments just below the cathode. The stimulus intensities will be adjusted for each testing condition, i.e. supine and sitting conditions. MMRs will be recorded bilaterally from hand and arm muscles and the trunk using low-noise, pre-amplified surface electromyographic electrodes placed on the skin over the muscle to record signal
Capabilities of Upper Extremity Questionnaire (CUE-Q) | From enrollment to the end of treatment at 4 weeks
  The Capabilities of Upper Extremity Questionnaire (CUE-Q) is designed to assess functional capabilities of the upper extremities, specifically in individuals that have experienced a neurological injury. The CUE-Q is a 32-item questionnaire, scored by self-report through an interview with the participant. The 32 items assess six domains including unilateral (left and right) items, bilateral items, reaching items, pulling/pushing items, wrist items, and hand and finger items.
Spinal Cord Injury-Quality of Life (SCI-QOL) Questionnaire | From enrollment to the end of treatment at 4 weeks
  The SCI-QOL was developed to address the shortage of psychometrically sound and relevant patient reported outcome measures available for clinical card and research in SCI rehabilitation. This questionnaire is accessible through computer adaptive testing and addresses the following domains: emotional health, physical-medical health, social participation, and physical function.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) - ASIA Impairment Scale (AIS) | From enrollment to the end of treatment at 4 weeks
  The ASIA Impairment Scale (AIS) is the most accepted classification in SCI that describes the level and severity of the injury, based upon the motor and sensory examination as described in the ISNCSCI for SCI. A "motor complete" injury (AIS A and B) is defined as an individual without motor sacral sparing (voluntary anal contraction) or sensory sacral sparing with motor function more than 3 levels below the motor level on either side. Motor incomplete injuries (AIS C and D) indicate some degree of sacral sparing and usually have voluntary movement in the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Forrest, Ph.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma P, Naglah A, Aslan S, Khalifa F, El-Baz A, Harkema S, D'Amico J. Preservation of functional descending input to paralyzed upper extremity muscles in motor complete cervical spinal cord injury. Clin Neurophysiol. 2023 Jun;150:56-68. doi: 10.1016/j.clinph.2023.03.003. Epub 2023 Mar 17. PMID 37004296
- [Background] Singh G, Sharma P, Forrest G, Harkema S, Behrman A, Gerasimenko Y. Spinal Cord Transcutaneous Stimulation in Cervical Spinal Cord Injury: A Review Examining Upper Extremity Neuromotor Control, Recovery Mechanisms, and Future Directions. J Neurotrauma. 2024 Sep;41(17-18):2056-2074. doi: 10.1089/neu.2023.0438. Epub 2024 Jul 12. PMID 38874496
- [Background] Sharma P, Panta T, Ugiliweneza B, Bert RJ, Gerasimenko Y, Forrest G, Harkema S. Multi-Site Spinal Cord Transcutaneous Stimulation Facilitates Upper Limb Sensory and Motor Recovery in Severe Cervical Spinal Cord Injury: A Case Study. J Clin Med. 2023 Jun 30;12(13):4416. doi: 10.3390/jcm12134416. PMID 37445450
- [Background] Zhang F, Momeni K, Ramanujam A, Ravi M, Carnahan J, Kirshblum S, Forrest GF. Cervical Spinal Cord Transcutaneous Stimulation Improves Upper Extremity and Hand Function in People With Complete Tetraplegia: A Case Study. IEEE Trans Neural Syst Rehabil Eng. 2020 Dec;28(12):3167-3174. doi: 10.1109/TNSRE.2020.3048592. Epub 2021 Jan 28. PMID 33382659
- See also: Tim and Caroline Reynolds Center for Spinal Stimulation at Kessler Foundation — https://kesslerfoundation.org/research/tim-and-caroline-reynolds-center-spinal-stimulation